CLINICAL TRIAL: NCT05961098
Title: A Phase II Clinical Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of RBD1016 Injection in Participants With Chronic Hepatitis B
Brief Title: A Study of RBD1016 in CHB Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Ribo Life Science Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RBHB1203
Record Dates: First submitted 2023-07-06; First posted 2023-07-27 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RBD1016/placebo 100 mg Q4W group (Experimental): Participants in the 100 mg Q4W dose group will receive corresponding doses of RBD1016 injection or placebo by subcutaneous injection on D1, D29, D57, and D85.
  Interventions: Drug: RBD1016
- RBD1016/placebo 200 mg Q4W group (Experimental): Participants in the 200 mg Q4W dose group will receive corresponding doses of RBD1016 injection or placebo by subcutaneous injection on D1, D29, D57, and D85.
  Interventions: Drug: RBD1016
- RBD1016/placebo 200 mg Q12W group (Experimental): Participants in the 200 mg Q12W dose group will receive corresponding doses of RBD1016 injection or placebo by subcutaneous injection on D1, and D85.
  Interventions: Drug: RBD1016

INTERVENTIONS:
Drug: RBD1016 — RBD1016 with NAs background treatment will be explored.

SUMMARY:
This study is a multi-center, randomized, double-blind, placebo-controlled clinical study to assess the safety, efficacy, PK and immunogenicity of RBD1016 injection on NAs background treatment in CHB participants.

DETAILED DESCRIPTION:
The study consists of screening period, treatment period, and FU period. It is divided into 3 dose groups, namely 100 mg Q4W, 200 mg Q4W and 200 mg Q12W. Each group will enroll 16 eligible participants, with 12 participants receiving RBD1016 injection and 4 participants receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for study participation;
2. Male or female participants aged 18-65 years;
3. Body mass index (BMI) within the range of 18-34 kilograms/square meter (kg/m2);
4. Documented history of chronic hepatitis B virus (HBV) infection, by positive HBsAg and/or HBV DNA tests ≥ 6 months before screening;
5. HBeAg positive or negative at screening;
6. On a stable regimen (≥ 12 months before screening) of any approved first-line oral NAs;
7. HBV DNA level <100 IU/mL at screening;
8. HBsAg level ≥50 IU/mL at screening;
9. Serum alanine aminotransferase (ALT) ≤ 1.5 times the upper limit of normal (ULN);
10. Liver transient elastography (FibroScan) results within 12 months before screening or at screening showing that the liver stiffness measurement (LSM) level is less than 9 kPa; or with liver biopsy within 24 months before screening showing that the Metavir score is F0-F2;

Exclusion Criteria:

1. Diagnosed with other liver diseases other than hepatitis B;
2. History of liver cirrhosis or hepatic decompensation (e.g., ascites, varices bleeding, or hepatic encephalopathy) before or at screening;
3. History of organ transplantation or previous or concurrent with hepatocellular carcinoma (HCC), or imaging findings suggesting a possibility of malignant liver lesions;
4. Concurrent hepatitis C virus (HCV), human immunodeficiency virus (HIV), or diagnosis of syphilis, acute hepatitis A or acute hepatitis E;
5. Laboratory results at screening as follows: serum alpha-fetoprotein (AFP) >50 μg/L; serum albumin concentration <3.0 g/dL; international normalized ratio (INR) >1.5; platelet count <90×10^9/L; serum direct bilirubin (DB) >2×ULN; serum creatinine concentration >1.5×ULN or creatinine clearance <60 mL/min (according to the Cockcroft-Gault equation); or any clinically significant laboratory outliers that the investigator believes may interfere with the interpretation of the efficacy and safety data in this study;
6. Those who the investigator believes are not suitable to participate in the study due to other factors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
safety: number and percentage of AEs | 24 weeks
  Number and percentage of participants with adverse events (AEs). All reported AE terms will be coded using Medical Dictionary for Drug Regulatory Affairs (MedDRA).
efficacy: the maximum decline of HBsAg level | 24 weeks
  The maximum decline (log value) of HBsAg level. Electro chmiluminescence method will be used to detect hepatitis B surface antigen (HBsAg).

SECONDARY OUTCOMES:
efficacy: the proportion of HBsAg decline≥1 log10 IU/mL | 24 weeks
  The proportion of participants with HBsAg decline ≥1 log10 IU/mL. Electro chmiluminescence method will be used to detect HBsAg.
PK parameter Cmax | 12 weeks
  Maximum concentration (Cmax) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
PK parameter Tmax | 12 weeks
  Time to maximum concentration (Tmax) will be calculated by PhoenixWinNonlin software (V8.0 or higher) will be used to calculate the PK parameter.
PK parameter AUC0-t | 12 weeks
  Area under the concentration-time curve from 0 to the collection time t (AUC0-t) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
PK parameter t1/2 | 12 weeks
  Half-Life (t1/2) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
PK parameter Vd/F | 12 weeks
  Apparent volume of distribution (Vd/F) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
PK parameter CL/F | 12 weeks
  Clearance (CL/F) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
PK parameter Css | 12 weeks
  Steady state concentration (Css) will be calculated by PhoenixWinNonlin software (V8.0 or higher).

CONTACTS AND LOCATIONS:
Locations (4):
- China (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Sweden (2):
  - Karolinska University Hospital, Stockholm, Stockholm County
  - Clinical Trial Consultants AB, Uppsala, Uppsala County

IPD SHARING:
Plan to Share IPD: No